CLINICAL TRIAL: NCT03858790
Title: Spinal Cord Stimulation System in the Treatment of Chronic Pain
Brief Title: Efficacy and Safety of Spinal Cord Stimulation in Patients With Chronic Intractable Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PINS-030
Record Dates: First submitted 2019-02-20; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pain; Chronic Pain; Back Pain; Spinal Cord Stimulation; Nervous System Diseases
Keywords: Pain
MeSH Terms: conditions — Pain; Chronic Pain; Back Pain; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects' PINS spinal cord stimulator randomized to this arm is on always
  Interventions: Device: PINS Spinal Cord Stimulator
- Control (Sham Comparator): Subjects' PINS spinal cord stimulator randomized to this arm is off for a week
  Interventions: Device: PINS Spinal Cord Stimulator

INTERVENTIONS:
Device: PINS Spinal Cord Stimulator — Subjects will be implanted with PINS spinal cord stimulator

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of spinal cord stimulation (SCS) using the PINS spinal cord stimulator device for chronic and intractable pain.

DETAILED DESCRIPTION:
Adult patients with chronic intractable pain of the trunk and/or limbs who are candidates for a treatment with spinal cord stimulation will be prospectively randomized into 2 arms. Spinal cord stimulation parameters are programmed and adjusted during outpatient clinic visits, within the normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with chronic, intractable pain of the trunk and/or limbs which has been refractory to conservative therapy for a minimum of 3 months.
2. VAS ≥ 5
3. Be 18 years of age or older at the time of enrollment
4. Be willing and able to comply with study-related requirements, procedures, and visits
5. Be willing and capable of giving informed consent

Exclusion Criteria:

1. Pregnancy or potential for with unwillingness to use contraception
2. Have a current diagnosis of a coagulation disorder, bleeding diathesis
3. Have evidence of psychiatric or cognitive disorder, who are unable to cooperate with surgery and program control
4. Have a life expectancy of less than 1 year
5. Have a condition currently requiring or likely to require the use of diathermy
6. Other inappropriate situations determined by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The difference of Visual-analogue scale (VAS) between the experimental group and the control group | 13 weeks
  Pain will be evaluated in the different groups according to the Visual-analogue scale (VAS) varying from 0 to 10 with a higher score indicating a higher level of pain.

SECONDARY OUTCOMES:
Changes in VAS | 4、12、24 weeks
  Pain will be evaluated in the different groups according to the Visual-analogue scale (VAS) varying from 0 to 10 with a higher score indicating a higher level of pain.
Sleep Quality | 4、12、24 weeks
  Quality of sleep will be assessed according to the number of nights with awakenings.
Changes in Beck Depression Inventory | 4、12、24 weeks
  This will be assessed using the Beck Depression Inventory, a self-report measure of depression severity that is a well-characterized scale with excellent psychometric properties and is frequently used in research studies of depression. Higher values represent greater severity of depression.
Change in quality of life as measured by SF-36 | 4、12、24 weeks
  The quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36) questionnaire.
Number of subjects with adverse events | 24 weeks
  The number of adverse events will be record at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] Lu Y, Xie D, Zhang X, Dong S, Zhang H, Yu B, Wang G, Wang JJ, Li L. Management of Intractable Pain in Patients With Implanted Spinal Cord Stimulation Devices During the COVID-19 Pandemic Using a Remote and Wireless Programming System. Front Neurosci. 2020 Dec 8;14:594696. doi: 10.3389/fnins.2020.594696. eCollection 2020. PMID 33363453
- [Derived] Lu Y, Mao P, Wang G, Tao W, Xiong D, Ma K, Li R, Feng D, Duan W, Li S, Fu Z, Feng Z, Jin Y, Wan L, Lu Y, Zhang D, Fan B, Wang JJ, Li L. Spinal cord stimulation for chronic intractable trunk or limb pain: study protocol for a Chinese multicenter randomized withdrawal trial (CITRIP study). Trials. 2020 Oct 7;21(1):834. doi: 10.1186/s13063-020-04768-3. PMID 33028415